CLINICAL TRIAL: NCT06602206
Title: Effects of Shoulder and Neck Mobilization on Pain, Sensation and Functionality in Patients With Subacromial Impingement Syndrome
Brief Title: Shoulder and Neck Mobilization in Patients With Subacromial Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06-29
Record Dates: First submitted 2024-07-30; First posted 2024-09-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional treatment group (Active Comparator): Hot packs, TENS, ultrasound, and exercise
  Interventions: Other: Conventional Treatment
- Conventional treatment + shoulder mobilization group (Experimental): Hot packs, TENS, ultrasound, exercise, and shoulder mobilization
  Interventions: Other: Conventional Treatment; Other: shoulder mobilization
- Conventional treatment + shoulder mobilization + neck mobilization group (Experimental): Hot packs, TENS, ultrasound, exercise, and shoulder and neck mobilization
  Interventions: Other: Conventional Treatment; Other: shoulder mobilization; Other: neck mobilization

INTERVENTIONS:
Other: Conventional Treatment — Hot pack,TENS, ultrasound and exercises
Other: shoulder mobilization — In the glenohumeral joint mobilization technique, distraction, anterior-posterior gliding, and inferior gliding movements will be applied.
  Arms: Conventional treatment + shoulder mobilization + neck mobilization group; Conventional treatment + shoulder mobilization group
Other: neck mobilization — Bridge, lateral flexion movement combined with traction, anterior-posterior gliding with traction, and lateral gliding techniques will be applied in neck mobilization.
  Arms: Conventional treatment + shoulder mobilization + neck mobilization group

SUMMARY:
Patients who come to Tavşanlı State Hospital's Physical Therapy and Rehabilitation Department and have been diagnosed with subacromial impingement syndrome by a physician will be included. Patients will be selected by randomization method among the patients determined by the physician to receive conservative treatment, shoulder mobilization in addition to conservative treatment, and neck mobilization treatment program in addition to these. Conventional treatments such as hot packs, TENS, ultrasound, and exercise will be given to all patients by the hospital staff. Pain intensity will be evaluated with VAS. Additionally, painful arch and pain-free joint range of motion evaluation will be made using a goniometer. The DASH questionnaire will be used to evaluate shoulder functionality. Sensory evaluation will be made with pressure pain threshold and two-point discrimination tests. Measurements will be made before the intervention and repeated after 3 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Diagnosed with Subacromial Impingement
* Not having received any treatment for shoulder problems in the last 6 months
* The pain has been continuing for 3 months
* Initial pain must be 4 or higher on the Visual Analog Scale (VAS)

Exclusion Criteria:

* History of surgery in the shoulder, cervical and thoracic region
* Having a shoulder problem such as a frozen shoulder or instability
* Full-thickness rotator cuff tear
* Having systemic musculoskeletal disease
* Having systemic rheumatic disease
* History of upper extremity fracture
* Diagnosed with scoliosis
* Have neurological problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | through study completion, an average of 1 year
  Pain intensity will be evaluated with VAS. VAS is a valid and reliable self-report scale consisting of a 10 cm long horizontal line, with scores ranging from 0 (no pain) to 10 (worst pain imaginable). Participants are asked to report the maximum pain they experienced in the last 24 hours. A change of 1.5 points is considered a minimal clinically important difference (MCID) for the VAS.

SECONDARY OUTCOMES:
The Arm, Shoulder and Hand Problems (DASH) Questionnaire | through study completion, an average of 1 year
  (DASH) questionnaire is a questionnaire that evaluates the functional level and disability of the entire upper extremity. At least 27 out of 30 questions must be answered for the inquiry to be evaluated. The query gives a value between 0-100. All questions are scored from 1 to 5. A higher score indicates greater disability.
Painful arch assessment | through study completion, an average of 1 year
  The patient is asked to abduct his arm as much as he can while standing or sitting. The test is positive if the patient feels pain between 60-120° of elevation. The sensitivity of the painful arc test performed in CNS patients was found to be 53% and the specificity was 80%.
Painless range of motion assessment | through study completion, an average of 1 year
  Painless ROM evaluation will be performed in CNS patients due to the presence of a painful arch. Pain-free ROM evaluation includes flexion and abduction movements occurring in the frontal and sagittal planes. These movements are evaluated using a universal goniometer. The patient is asked to actively create 2 movements in a standing or sitting position. While performing measurements with a goniometer, the part with pain-free ROM will be noted in degrees
Pressure-pain Threshold Assessment | through study completion, an average of 1 year
  Pressure pain threshold is the most commonly used method among quantitative sensory tests.Measurements will be taken from the upper trapezius, supraspinatus, and middle deltoideus muscles.
Evaluation of Tactile Sensory Acuity | through study completion, an average of 1 year
  Esthesiometer measurements will be taken from the surfaces corresponding to the C5, C6, and C7 dermatomes. To standardize the test areas, vertical lines will be drawn from the anterior, middle, and posterior edges of the acromion towards the elbow. The test will begin at 0 mm and the distance will first be gradually increased in 5 mm increments until the participant perceives two dots instead of one. When the participant reports detecting two dots, that distance will be recorded. Separate evaluations will be taken from 3 regions and the results will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Işıntaş, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No